CLINICAL TRIAL: NCT01797679
Title: Efficacy of Strength and Aerobic Exercise on the Articular Cartilage of Patients With Mild and Moderate Knee Osteoarthritis Measured by T2 and T1 Rho MR Imaging - A Randomized Controlled Trial
Brief Title: Study of Cartilage Relaxometry and Physical Activity in Osteoarthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of agreement between the participants and lack og funding
Sponsor: University Hospital, Akershus (Other)
Collaborators: The Research Council of Norway (Other); Oslo University Hospital (Other); Hjelp24 (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Hasan Banitalebi, Radiologist, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NFR213335/h10
Record Dates: First submitted 2013-02-21; First posted 2013-02-22 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis,Articular Cartilage, Relaxometry, Morphometry, MRI, T2 mapping, T1 rho
MeSH Terms: conditions — Osteoarthritis | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Strength Training (Other): The strength group include progressive strength training and neuromuscular exercises. The inclusion will be performed 2-3 times a week for 12 weeks.
  Intervention: Other: Strength training
  Interventions: Other: Strength Training
- Aerobic exercise (Experimental): The aerobic exercise group will cycle on an ergometer bicycle 2-3 times a week for 12 weeks on moderate loading. The loading will be controlled by a heart rate monitor and is defined as 85% of maximal heart rate.
  Interventions: Other: Aerobic Exercise
- Control Group (No Intervention): The control group will do as usual.

INTERVENTIONS:
Other: Strength Training
  Arms: Strength Training
Other: Aerobic Exercise
  Arms: Aerobic exercise

SUMMARY:
This study is the radiological component of an earlier registered trial under the title: Efficacy of Exercise on Physical Function and Cartilage Health in Patients With Knee Osteoarthritis. The main purpose in this component of the study is to evaluate the efficacy of aerobic exercise and strength training on the T2 and T1 rho relaxation times of the articular cartilage. It has been proven that exercise can improve function and reduce the need for analgesics in patients with osteoarthritis. With this study, we wish to investigate if different kinds of exercise can cause measurable improvements in T2 and T1 rho relaxation times of the articular cartilage, and also if this improvements are transient or permanent.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 45-65 years
* Clinical knee OA according to the American College of Rheumatology Clinical Criteria 17
* Kellgren and Lawrence radiographic OA grade 2 and 3 (mild to moderate radiographic OA)

Exclusion Criteria:

* Severe knee OA according to the Kellgren and Lawrence classification (grade 4)
* Other known major musculoskeletal impairments in the lower extremities or the back or prostheses in any joint of the lower extremities
* Known coronary heart diseases or cancer
* Body mass index > 35
* Scheduled for surgery in any joint
* Known mental or psychologic diseases
* Known drug abuse
* Persons who already perform sports related moderate physical activity more than two times a week
* Contraindications for magnetic resonance imaging (specific point list at Diagnostic Imaging Division, Akershus University Hospital)
* Not speaking Norwegian

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Qualitative Cartilage Morphology Assessment | One year
  Indirect cartilage morphology will by assessed by X-ray Direct cartilage morphology will be assessed by MRI morphometry The biochemical composition of the cartilage will be assessed by relaxometry (T2 and T1 rho relaxation times)

SECONDARY OUTCOMES:
Semiquantitative Cartilage Assessment | One year
  Using semiquantitative techniques, the clinical manifestations of osteoarthritis assessed by MRI such as: cartilage lesions and bone marrow lesions will be assessed and quantified by MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Lorenskog, Norway

IPD SHARING:
Plan to Share IPD: No